CLINICAL TRIAL: NCT02797574
Title: Stress Response Pathways in Vitiligo: A Prospective, Investigator Initiated, Interventional Study With Two Arms
Brief Title: Stress Response Pathways in Vitiligo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-00445
Record Dates: First submitted 2016-02-04; First posted 2016-06-13 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitiligo Diagnosed Group (Active Comparator): Clinically diagnosed with non-segmental vitiligo
  Interventions: Procedure: Punch Biopsy at a Lesional Site; Procedure: Punch Biopsy at a Non- Lesional site
- Healthy Control Group (Active Comparator): 20 normally pigmented control subjects who are between the ages of 18 and 50
  Interventions: Procedure: Punch Biopsy at a Non- Lesional site

INTERVENTIONS:
Procedure: Punch Biopsy at a Lesional Site
  Arms: Vitiligo Diagnosed Group
Procedure: Punch Biopsy at a Non- Lesional site

SUMMARY:
The purpose of this study is to investigate stress response pathways in tissues and melanocytes from patients with vitiligo. Investigators are collecting evidence of UPR and stress response activation in tissues and melanocytes from patients with vitiligo. Individuals with vitiligo will have punch biopsies to study stress response UPR activation and NF-κB signaling to test our hypothesis. In order to characterize differences between disease and normal states, a second arm of control individuals (Arm 2) will be recruited.

DETAILED DESCRIPTION:
Identifying a role for NF-κB signaling in vitiligo may improve therapies for this disfiguring disorder. Current treatments vary in effectiveness and may not always be long lasting cases. The NF-κB pathway and IL-6 itself are the target of several FDA approved drugs, thus opening new therapeutic avenues.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for participation, subjects must meet all of the following criteria:
* Must have a clinical exam consistent with and diagnosis of non-segmental vitiligo
* Must be normally pigmented
* No clinical presentation of vitiligo

Exclusion Criteria:

* Outside of the specified age range
* No clinical diagnosis of vitiligo
* Use of systemic therapies, including but not limited to methotrexate, etretinate, or cyclosporine, calcineurin inhibitors and/ or vitamin D analogs within 4 weeks of enrollment
* Use of topical steroids or topical immunodilators at biopsy site within 4 weeks of enrollment
* History of keloids or hypertrophic scars
* Patients with pacemakers or defibrillators or heart valves
* Patients on Plavix, Warfarin or similar anticoagulation medicine
* Pregnant females
* Lactating women
* Allergies or sensitivity to lidocaine or epinephrine
* Outside of the specified age range
* Abnormally pigmented at potential biopsy sites (non-vitiligo)
* Clinical presentation of vitiligo
* Use of systemic therapies, including but not limited to methotrexate, etretinate, or cyclosporine, calcineuron inhibitors and/ or vitamin D analogs within 4 weeks of enrollment
* Use of topical steroids or topical immunodilators at biopsy site within 4 weeks of enrollment
* History of keloids or hypertrophic scars

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
T-test measures of expression levels of target proteins in patients versus controls (p < 0.05) | 1 Year

SECONDARY OUTCOMES:
T-test measures of expression levels in response to Vitiligo triggers | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Prashiela Manga, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States